CLINICAL TRIAL: NCT06267599
Title: ACAR-Style Bladder Suture in Uterus-Sparing Surgery and Hysterectomy for Placenta Percreta: A Result Analysis
Brief Title: Bladder Suture in Uterus-Sparing Surgery and Hysterectomy for Placenta Percreta
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Cemre Alan, Fellow, Necmettin Erbakan University
Other Study IDs: ACAR-Style Bladder Suture
Record Dates: First submitted 2024-01-15; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Placenta Percreta; Bladder Injury; Sutures
Keywords: Placenta Percreta, Bladder Invasion, Sutures
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bladder suture group: This group consisted of patients in whom we could not open the bladder and uterine cervix by dissection, so we had to open the bladder. In this group, the bladder dome was opened and a special suture was passed through the bladder to control bleeding. This procedure was performed to control bleeding.
  Interventions: Procedure: ACAR-Style Bladder Suture
- Control group: For the patients in this group, the vascular structures between the bladder and cervix were coagulated one by one. The bladder was not opened during this procedure.

INTERVENTIONS:
Procedure: ACAR-Style Bladder Suture — In cases where dissection is not possible, the upper border of the bladder is opened transversely with a cutter, and the ureteral catheters and trigone inside the bladder are observed. The bladder invasion border is re-evaluated intravesically. The uterine arteries are held bilaterally with a sensitive clamp that does not crush the uterine arteries. Then, the uterus is incised from the upper border of the bladder without damaging the bladder and the predetermined myometrial invasion area is resected. After the placenta is removed, the cervical canal is found and marked with a number one vicryl suture. In these patients, the placental material is removed in pieces in the cervix area where the bladder is invaded. After the removal of the placenta, the cervix in the lower segment of the uterus is orientated and sutured together with the bladder, and this area is closed.
  Groups: Bladder suture group

SUMMARY:
This study aimed to evaluate the short-term and long-term complications of placenta percreta with bladder invasion. This evaluation focuses on cases where bladder dissection and ACAR-style bladder sutures were applied in cases of placenta percreta with bladder invasion that underwent uterine-sparing surgery or hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Clinical diagnosis of PAS
* PAS with bladder invasion

Exclusion Criteria:

* Cases with incomplete or inadequate medical records
* Cases with other types of placental invasion (e.g., placenta accreta, placenta increta),
* Cases with missing key data points.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women who underwent surgery for PAS and bladder invasion between January 2018 and January 2023 in a tertiary university hospital in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Comparison of intraoperative bleeding and complication rates of the two groups | during operation time
  It was observed that the amount of intraoperative bleeding (volume aspirated cc blood), surgical time (minutes), blood transfusion rates (%), and hysterectomy rates(%).
Comparison of postoperative bleeding between two groups | postoperative three days,
  It was observed that the amount of postoperative bleeding (hemoglobin(g/dL) change, need for blood transfusion Unite)
Comparison of complication rate between two groups | six months postoperatively
  It was described as long-term bladder dysfunction(Nocturia, Urgency, Stress urinary incontinance, fistula rate (%))
  Nocturia: Waking up more than once during the night. Urgency: Sudden, intense urge to urinate followed by an involuntary loss of urine.
  Stress urinary incontinance: Happens when physical movement or activity - such as coughing, laughing, sneezing, running or heavy lifting - puts pressure (stress) on your bladder, causing you to leak urine.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Acar, Study Director — MD; Şükran Doğru, Principal Investigator — MD; Fatih Akkuş, Study Chair — MD; Cemre Alan, Study Chair — MD; Fikriye Karanfil Yaman, Study Chair — MD; Huriye Ezveci, Study Chair — MD; Orhan Ay, Study Chair — MD; Fethiye Şahin, Study Chair — MD; Burçin Elaziz, Study Chair — MD; Meryem Gümüş, Study Chair — MD
Locations (1):
- Cemre Alan, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Horgan R, Hessami K, Hage Diab Y, Scaglione M, D'Antonio F, Kanaan C, Erfani H, Abuhamad A, Shamshirsaz AA. Prophylactic ureteral stent placement for the prevention of genitourinary tract injury during hysterectomy for placenta accreta spectrum: systematic review and meta-analysis. Am J Obstet Gynecol MFM. 2023 Oct;5(10):101120. doi: 10.1016/j.ajogmf.2023.101120. Epub 2023 Aug 5. PMID 37549736
- [Background] Couret M, Huang Y, Khoury-Collado F, Friedman A, Hou JY, St Clair CM, Tergas AI, Ananth CV, Wright JD. Patterns of care for women with placenta accreta spectrum. J Matern Fetal Neonatal Med. 2021 Oct;34(20):3370-3376. doi: 10.1080/14767058.2019.1684471. Epub 2019 Nov 19. PMID 31744356
- [Background] Committee on Obstetric Practice. Committee opinion no. 529: placenta accreta. Obstet Gynecol. 2012 Jul;120(1):207-11. doi: 10.1097/AOG.0b013e318262e340. PMID 22914422
- [Background] Society of Gynecologic Oncology; American College of Obstetricians and Gynecologists and the Society for Maternal-Fetal Medicine; Cahill AG, Beigi R, Heine RP, Silver RM, Wax JR. Placenta Accreta Spectrum. Am J Obstet Gynecol. 2018 Dec;219(6):B2-B16. doi: 10.1016/j.ajog.2018.09.042. PMID 30471891
- [Background] Woldu SL, Ordonez MA, Devine PC, Wright JD. Urologic considerations of placenta accreta: a contemporary tertiary care institutional experience. Urol Int. 2014;93(1):74-9. doi: 10.1159/000356064. Epub 2014 Apr 9. PMID 24732915
- [Background] Erfani H, Salmanian B, Fox KA, Coburn M, Meshinchiasl N, Shamshirsaz AA, Kopkin R, Gogia S, Patel K, Jackson J, Cadena M, Aalipour S, Sukumar S, Nassr AA, Espinoza J, Clark SL, Belfort MA, Shamshirsaz AA. Urologic morbidity associated with placenta accreta spectrum surgeries: single-center experience with a multidisciplinary team. Am J Obstet Gynecol. 2022 Feb;226(2):245.e1-245.e5. doi: 10.1016/j.ajog.2021.08.010. Epub 2021 Aug 13. PMID 34391750
- [Background] Wu WJ, Smith AD, Okeke Z. Bladder Necrosis Associated with Placenta Accreta, Embolization, and Repair of Cystotomies. J Endourol Case Rep. 2015 Oct 1;1(1):24-6. doi: 10.1089/cren.2015.29007.wjw. eCollection 2015. PMID 27579379
- [Background] Li GT, Li XF, Ding Y. Cervicovesical U-suture: An effective novel alternative to partial cystectomy for controlling life-threatening postpartum hemorrhage due to placenta accreta spectrum invading the bladder. Asian J Surg. 2022 Dec;45(12):2745-2747. doi: 10.1016/j.asjsur.2022.06.018. Epub 2022 Jun 18. No abstract available. PMID 35729022
- [Background] Acar A, Ercan F, Pekin A, Elci Atilgan A, Sayal HB, Balci O, Gorkemli H. Conservative management of placental invasion anomalies with an intracavitary suture technique. Int J Gynaecol Obstet. 2018 Nov;143(2):184-190. doi: 10.1002/ijgo.12593. Epub 2018 Aug 13. PMID 29989156
- [Background] Feng JP, Fan DZ, Lin DX, Zhang HS, Rao JM, Liu ZP. Sandwich excision in patients with placenta percreta involving maternal bladder. Eur Rev Med Pharmacol Sci. 2022 Jun;26(12):4252-4257. doi: 10.26355/eurrev_202206_29062. PMID 35776024
- [Background] Matsuzaki S, Yoshino K, Endo M, Kakigano A, Takiuchi T, Kimura T. Conservative management of placenta percreta. Int J Gynaecol Obstet. 2018 Mar;140(3):299-306. doi: 10.1002/ijgo.12411. Epub 2018 Jan 3. PMID 29194646
- [Background] Matsubara S. Intentional cystotomy in surgery for placenta percreta with bladder invasion: Not only for hysterectomy but also for uterus-preserving surgery. Acta Obstet Gynecol Scand. 2023 Jan;102(1):122-123. doi: 10.1111/aogs.14484. Epub 2022 Nov 30. No abstract available. PMID 36448372
- [Background] Scaglione MA, Allshouse AA, Canfield DR, Mclaughlin HD, Bruno AM, Hammad IA, Branch DW, Maurer KA, Dood RL, Debbink MP, Silver RM, Einerson BD. Prophylactic Ureteral Stent Placement and Urinary Injury During Hysterectomy for Placenta Accreta Spectrum. Obstet Gynecol. 2022 Nov 1;140(5):806-811. doi: 10.1097/AOG.0000000000004957. Epub 2022 Oct 5. PMID 36201777
- [Background] Matsubara S, Takahashi H, Baba Y. Handling aberrant vessels located in the posterior bladder wall in surgery for abnormally invasive placenta: a non/less-touch technique. Arch Gynecol Obstet. 2017 Nov;296(5):851-853. doi: 10.1007/s00404-017-4498-2. Epub 2017 Sep 5. PMID 28875376
- [Background] Friedrich L, Mor N, Weissmann-Brenner A, Kassif E, Friedrich SN, Weissbach T, Castel E, Levin G, Meyer R. Risk factors for bladder injury during placenta accreta spectrum surgery. Int J Gynaecol Obstet. 2023 Jun;161(3):911-919. doi: 10.1002/ijgo.14567. Epub 2022 Nov 28. PMID 36353748
- [Background] Crocetto F, Saccone G, Raffone A, Travaglino A, Gragnano E, Bada M, Barone B, Creta M, Zullo F, Imbimbo C. Urinary Incontinence after Planned Cesarean Hysterectomy for Placenta Accreta. Urol Int. 2021;105(11-12):1099-1103. doi: 10.1159/000518114. Epub 2021 Aug 18. PMID 34515253
- See also: Dogru S, Akkus F, Atci AA et al. (2022) The fetal and maternal outcomes related to previous number of cesarean sections and uterus sparing surgery in women with abnormal placentation. Journal of Clinical and Investigative Surgery 7:29-30. — https://doi.org/10.25083/2559.5555/7.1.5
- See also: Doğru Ş, Altınordu Atcı A, Akkuş F et al. (2022) Use of ureteral catheter in uterine-sparing surgery for placenta accreta. Perinatal Journal 30:158-164. — https://doi.org/10.2399/prn.22.0302009